CLINICAL TRIAL: NCT04510064
Title: Conversion Effects of PD-1 Antibody Camrelizumab Combined With Nab-POF Regimen Chemotherpy in Patients With Initially Unresectable Locally Advanced or Limited Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma：FDZL-GC001 Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-PFG
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Gastric Cancer; Locally Advanced Gastric Adenocarcinoma; Gastric Cancer Adenocarcinoma Metastatic
Keywords: gastric cancer; gastroesophageal adenocarcnoma; conversion chemotherapy; PD-1antibody
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: Patients were treated with domestic PD-1 antibody (Camrelizumab for injection) commbined with mFLOT regimen, and HER-2 positive patients were added Herceptin therapy. If primary tumor and metastatic lesions could be converted to R0 resection after 6-9 cycles of immunochemotherapy, then proceeded to surgery,otherwize treated according to the principles of palliative care. Patiens after surgery continued prior immunotherapy to 12 cycles or intolerable toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients were treated with domestic PD-1 antibody (Camrelizumab for injection) commbined with mFLOT regimen immunotherapy every two weeks, and HER-2 positive patients were added with Herceptin therapy. Camrelizumab 200mg on day 1, albumin bound paclitaxol 125mg/m² on day 1,oxaliplatin 85 mg/m² on day 1, leucovorin 200 mg/m² on day 1, and 5-FU 2600 mg/m² as 24-h infusion on day 1.Herceptin 6mg/Kg at the first time, followed by 4mg/Kg if needed.The efficacy of therapy was evaluated every 3 treatment cycles. If the tumor can be R0 resected after 6-9 cycles, then proceeded to surgery. After the operation, patients continued to receive the prior immunotherapy totally to 12 cycles or to the disease progressed or intolerable toxicity.
  Interventions: Drug: Camrelizumab plus mFLOT regimen; Procedure: R0 surgery

INTERVENTIONS:
Drug: Camrelizumab plus mFLOT regimen — Patients were treated with domestic PD-1 antibody (Camrelizumab for injection) commbined with mFLOT regimen immunotherapy every three weeks, and HER-2 positive patients were added with Herceptin therapy. Camrelizumab 200mg on day 1, albumin bound paclitaxol 125mg/m² on day 1,oxaliplatin 85 mg/m² on day 1, leucovorin 200 mg/m² on day 1, and 5-FU 2600 mg/m² as 24-h infusion on day 1.Herceptin 6mg/Kg at the first time, followed by 4mg/Kg if needed.
Procedure: R0 surgery — The efficacy of therapy was evaluated every 3 treatment cycles. If the tumor can be R0 resected after 6-9 cycles, then proceeded to surgery. After the operation, patients continued to receive the prior immunotherapy totally to 12 cycles or to the disease progressed or intolerable toxicity.

SUMMARY:
This study is to evaluate the efficacy and safety of domestic programmed death 1（ PD-1） antibody (Camrelizumab for injection) combined with fluorouracil plus leucovorin, oxaliplatin, and albumin bound paclitaxel (Nab-POF) regimen in the treatment of patients with unresectable locally advanced or limited metastatic gastric cancer. The primary efficacy endpoint is R0 resection rate.

DETAILED DESCRIPTION:
This is an open, single center, prospective phase II clinical study to evaluate the efficacy and safety of domestic PD1 antibody (Camrelizumab for injection) combined with Nab-POF regimen in the treatment of unresectable locally advanced or limited metastatic gastric cancer. This study will be carried out in our center, about 40 patients will be enrolled.

Patients with unresectable locally advanced or limited metastatic gastric cancer who had not received any prior antitumor therapies were treated with domestic PD1 antibody (Caerelizumab for injection) commbined with mFLOT regimen, and human epidermal-growth-factor receptor 2 (HER-2) positive patients were treated with Herceptin. The efficacy of therapy was evaluated every 3 treatment cycles. After 6 cycles, surgical experts evaluated the resectability of the tumor, and the patients who were confirmed to be resectable received surgery within 3-6 weeks after immunochemotherapy. The patients with good postoperative recovery continued to receive the same immunochemotherapy in 3-6 weeks, and totally at most 12 cycles. Patients who were evaluated as progressive disease (PD) at any time withdrawn from the study as conversion failure.Patients who did not PD at 6 cycles of treatment but did not reach the criteria for R0 resection, continued to receive another 3 cycles of the prior chemotherapy. If resectable then, surgical treatment was performed, if still unresectable, the immunochemotherapy for transformation was evaluated as unsuccessful. The patients were treated according to the principle of palliative treatment until the disease progressed or intolerable toxicity. The efficacy and safety will be continuously monitored and evaluated throughout the study period (including a 30 day follow-up period). 40 cases were expected to be enrolled: 3-4 cases per month, completed in 1 year and finished in 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry, no gender limit.
* Participants must have histologically or cytologically confirmed adenocarcinoma of the stomach (including adenocarcinoma of the gastroesophageal junction).
* At least one measurable site of disease as defined by RECIST criteria with spiral CT scan or MRI.
* CT or MRI showed unresectable locally advanced gastric cancer (imaging stage T4b and / or second station lymph node > 3cm or fusion mass) or limited metastatic gastric cancer with any of the following single site metastasis:

  1. Retro-peritoneal lymph node metastasis (RPLM) (e.g. para-aortic, intra-aorto-caval, para-pancreatic or mesenteric lymph nodes).
  2. Single or bilateral Krukenberg tumors.
  3. No more than 5 liver metastases, and the maximum diameter of the lesions was less than 5 cm.
  4. Adrenal metastasis.
  5. Localized potentially operable peritoneal carcinomatosis: stage P1 according to classification of the"Japanese Research Society for Gastric Cancer (JRSCGC)".
* No clinically visible peritoneal metastasis (such as CT imaging confirmation or ascites).
* No prior anti-tumor therapy.
* Performance status (PS) < 2 (ECOG scale).
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: hemoglobin≥90g/dL,absolute neutrophil count ≥ 1.5×109/L, platelets ≥100 x109/L; Total bilirubin < 1.5x upper normal limit (UNL), Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) <2.5 x ULN, if liver metastasis existed, SGOT,SGPT<2.5xULN. International normalized ratio (INR) ≤2.5 x ULN, Serum Creatinine ≤ 1 x institutional ULN or creatinine clearance (CrCl) >50ml/min (if using the Cockcroft-Gault formula ).
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* A history of other malignancies within 3 years prior to enrollment, except for cervical carcinoma in situ or skin basal cell carcinoma that had been cured.
* Accompanied with brain or meningeal metastasis.
* Malignant pleural and peritoneal effusion.
* Accompanied by gastrointestinal obstruction, gastrointestinal bleeding (fecal occult blood +++ )or perforation.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137,or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has an active or history of autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or with high risk (such as receiving immunosuppressive therapy after organ transplantation), but in the past two years with vitiligo, psoriasis, alopecia or Graves' disease without systemic treatment, hypothyroidism with thyroid hormone replacement therapy only and type I diabetes only need insulin replacement therapy can be enrolled.
* Suffering from interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease and radiation pneumonia.
* Participate in other clinical studies of drugs (subject to the use of trial drugs) within 4 weeks before the first administration, unless participating in observational (non intervention) clinical studies.
* Used immunosuppressive drugs within 4 weeks before the first dose of study treatment, excluding nasal, inhalation or other local glucocorticoids or physiological doses of systemic glucocorticoids (i.e. no more than 10mg prednisone or equivalent dose of other glucocorticoids, or short-term (no more than 7 days) use of glucocorticoids to prevent or treat non autoimmune allergic diseases.
* Planned to receive live attenuated vaccine within 4 weeks before the first dose of study treatment or during the study period. Note: inactivated virus vaccine for seasonal influenza is allowed within 4 weeks before the first administration, however, live attenuated influenza vaccine is not allowed.
* Major surgery (craniotomy, thoracotomy or laparotomy) was performed within 4 weeks before the first dose of study treatment, or major surgery (not in this study) was expected to be performed during the study treatment.
* A history of HIV infection (i.e. HIV antibody positive), or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or stem cell transplantation.
* Patients with active chronic hepatitis B or active hepatitis C, hepatitis B virus carriers. Stable hepatitis B after drug treatment (DNA titer not higher than 200iu/ml or copy number < 1000copies / ml) and cured patients with hepatitis C (HCV RNA test negative) can be included in the group.
* Active tuberculosis.
* Severe infection within 4 weeks before the first administration, or active infection within the first 2 weeks and requiring oral or intravenous antibiotic treatment.
* Symptomatic congestive heart failure (NYHA grade II-IV) or symptomatic or poorly controlled arrhythmias;
* Uncontrolled arterial hypertension (systolic blood pressure≥160mmhg or diastolic blood pressure≥100mmhg) even after standard treatment.
* Any arterial thromboembolism events, including myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before the treatment.
* A history of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months before enrollment (implantable venous infusion port or catheter-derived thrombosis, or superficial venous thrombosis is not considered as "severe" thromboembolism)
* Have a clear history of neurological or mental disorders in the past, such as epilepsy, dementia, poor compliance, or patients with peripheral nervous system disorders.
* Alcohol addicts or have a history of drug use or drug abuse in the past 1 yea.
* Pregnant or lactating women, fertile women without adequate contraceptive measures
* Other acute or chronic diseases, mental disorders, or laboratory test value abnormalities that may result in increased risk associated with study participation or drug administration, or interference with the interpretation of the study results, and the patient, in the judgment of the investigator, is not eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
margin-free-(R0) resection rate | 6-9 weeks after immunochemotherapy
  R0 resection was defined as no tumor identified on microscopic examination of proximal, distal,or circumferential margins.

SECONDARY OUTCOMES:
pathological complete response (pCR) | 6-9 weeks after immunochemotherapy and R0 surgery
overall response rate (ORR) | up to 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 24 months
sugery complications | up to 2 months after the period of surgery
  sugery complications
progression free survival (PFS) | up to 24 months
  randomisation to disease progression, relapse, or death; surgical morbidity and mortality
overall survival (OS) | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: weijian guo, professor, Principal Investigator — Fudan university, Shanghai Cancer Certer
Locations (1):
- Fudan University, Shanghai Cancer Center, Shanghai, Shanghai Municipality, China